CLINICAL TRIAL: NCT05106608
Title: Photobiomodulation Therapy With M-health Tool for the Management of Oral Health and Quality of Life in Head and Neck Cancer Patients: LAXER Study
Brief Title: Photobiomodulation Therapy Plus M-health in Head and Neck Cancer Patients: LAXER Study
Acronym: LAXER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Noelia Galiano-Castillo, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBM_CANCER21; PI-0187-2021 (Other Grant/Funding Number: Conserjeria de Salud y Familias (Junta de Andalucía))
Record Dates: First submitted 2021-10-10; First posted 2021-11-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Xerostomia
Keywords: Quality of Life; Neoplasms; Xerostomia; Low-Level Light Therapy; Telemedicine
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants who meet the inclusion and exclusion criteria will be randomized to one of the three study groups using a random number generation program (www.randomizer.org). The randomization sequence will be prepared by a member external to the investigation to respect the masking in terms of randomization of the participants, thus reducing the risk of bias during the evaluations. Therefore both patients and evaluator will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group PBM_1 (Experimental): Energy density 7.5 J / cm2 for group PBM_1
  Interventions: Device: Energy density photobiomodulation (7.5)
- Group PBM_2 (Experimental): Energy density 3 J / cm2 for group PBM_2
  Interventions: Device: Energy density photobiomodulation (3)
- Placebo Control (Placebo Comparator): The placebo control group will carry out the same protocol used in irradiated patients (including the use of protective glasses) using the same laser device to imitate a real irradiation; however, the device will be turned off and a recording of the emission sounds will be used to give the patient the hearing sensation of the laser therapy.
  Interventions: Device: Sham placebo

INTERVENTIONS:
Device: Energy density photobiomodulation (7.5) — A total of 22 points will be treated (extraoral and intraoral). 2 sessions per week, for 3 months (24 sessions in total). In addition, a mobile health application (LAXER) will be provided.
  Arms: Group PBM_1
Device: Energy density photobiomodulation (3) — A total of 22 points will be treated (extraoral and intraoral). 2 sessions per week, for 3 months (24 sessions in total). In addition, a mobile health application (LAXER) will be provided.
  Arms: Group PBM_2
Device: Sham placebo — In addition, a mobile health application (LAXER) will be provided.
  Arms: Placebo Control

SUMMARY:
The Photobiomodulation therapy could have positive effects on quality of life and oral health in head and neck cancer survivors post-radiotherapy. The improvement in quality of life will be maintained after a follow-up period.

DETAILED DESCRIPTION:
Many experts advocate the use of Photobiomodulation (PBM) therapy in patients with cancer and demand studies of higher methodological quality such as randomized controlled clinical trials. However, there is no consensus on the most effective dosimetry that allows us to establish an effective and safe approach to treat radiotherapy-induced xerostomia in head and neck cancer survivors. Finally, recent reviews highlight the importance of determining whether or not the effects of Photobiomodulation therapy are maintained after a follow-up period.

ELIGIBILITY:
Patients will be included in the study if they meet the following inclusion criteria:

* men or women aged 18 years or older and were diagnosed with HNC.
* chronic xerostomia.
* received RT in the parotid, submandibular and/or sublingual salivary glands.
* grade 3 oral dryness according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE).
* medical treatment completed and in complete remission.
* received medical clearance for participation in this study.
* at least one month passed since the end of RT to avoid the possible presence of oral mucositis and/or radiodermatitis, which limits adherence to treatment and maximum 36 months.
* no history of drugs/devices/products (pilocarpine, cevimeline, amifostine, oral devices, humidifiers, or herbs) to prevent or treat xerostomia prior to study inclusion or no change in their use (no change in type or dose) for two months prior to study inclusion.
* and able to access mobile applications or living with someone who has this ability.

The exclusion criteria will be as follows:

* patients with metastases.
* a score <60 on the Karnofsky Performance Status Scale.
* contraindications to receiving PBM therapy (e.g., cardiac arrhythmias, pacemakers, photosensitivity, drugs with photosensitizing action, and pregnancy).
* other comorbidities such as diabetes and polypharmacy.
* and retraction of the declaration of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
General and specific quality of life. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 comprises 30 items on 5 functional scales, 3 symptom scales, 6 single items and a global health scale measured by a 4-point Likert scale with a total score ranging from 0 to 100. Higher scores on the functional and global health scales indicate better functioning or QoL, respectively, but higher scores on the symptom scales or single items indicate a high level of symptoms. In addition, the specific head and neck module (EORTC QLQ-H&N35) will be used; this module comprises 35 items on 7 multi-item scales and 11 single items scored from 0 to 100. Higher scores indicate more symptoms.
Oral Health. Severity of xerostomia. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  Xerostomia Inventory consists of 11 items (score range 1-5) with a total score ranging from 11 to 55 points to rate the severity of chronic xerostomia. A higher score indicates more severe xerostomia.
Oral Health. Dysphagia. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  Eating Assessment Tool questionnaire (EAT-10) consists of 10 items related to swallowing difficulties (score range 0-4, 0=no problem, 4=severe problem), with a total score of 3 or higher indicating dysphagia.
Oral Health. Perceived xerostomia. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  A numeric visual analog scale (VAS) will be used with with a grade ranging from 0 (no symptoms) to 10 (the worst possible symptoms).
Oral Health. Degree of mouth opening. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The degree of mouth opening will be determined by the range of motion (ROM) using a sliding caliper, which will measure the maximal interincisal distance in millimeters.
Oral Health. Clinical physical findings (dryness in the mouth). | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  A total of 10 examples of clinical physical findings where each one represents a feature of dryness in the mouth will be administered through the Clinical Oral Dryness Score (CODS). A score of 2 or more indicates significant oral dryness.
Oral Health. Regional oral dryness. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  Regional Oral Dryness Inventory (RODI) quantifies the severity of dryness at 9 different locations in the oral cavity and is represented by 9 illustrations. Patients will indicate the severity of perceived oral dryness using a 5-point Likert scale (1=none, 5=severe).
Salivary secretion. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The 5-min unstimulated and 5-min stimulated salivary flow rates (SFRs) will be calculated (ml/min) and the volume of each sample will be also calculated (in microlitres). Samples from unstimulated saliva will be used to analyse salivary biomarkers, such as proteins (e.g., antibodies), calcium concentration and pH, using commercial kits.
Salivary gland ultrasound assessment. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The morphology of the parotid and submandibular glands will be assessed using 2D echography (Samsung HM70A echograph) to quantify changes in size in three dimensions.

SECONDARY OUTCOMES:
Pressure pain threshold. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  An electronic algometer (SENSEBox System, Somedic AB, Sösdala, SE) will be used to assess pain at 7 body sites bilaterally: the C5-C6 joint, upper trapezius, elevator scapulae, masseter, temporalis, sternoclavicular joint and tibialis anterior distal point. The mean of the three measurements will be considered.
Functional Performance. Functional capacity. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The 6-minute walk test (6MWT) will be used; the maximum walked distance (meters) that patients are able to walk in a 30-meter linear corridor will be quantified. A longer distance indicates better functional capacity.
Functional Performance. Mobility/fall risk. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The timed up-and-go (TUG) test will be used; patients sit back in a chair and walk toward a cone located 3 meters away as quickly as possible. The time (seconds) needed will be registered 2 times, with a shorter time indicating better mobility.
Functional Performance. Perceived fitness status. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The International Fitness Scale (IFIS) assesses overall fitness, cardio-respiratory fitness, muscular strength, speed/agility and flexibility dimensions, using a 5-point Likert scale (1=very poor, 2=poor, 3=average, 4=good, 5=very good).
Functional Performance. Physical activity level. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The International Physical Activity Questionnaire Short Form (IPAQ-SF), a self-reported validated questionnaire in patients with cancer that records the activities of the previous 7 days according to intensity level.
Mood. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  The Spanish version of the Scale for Mood Assessment (EVEA) will also be used and comprises 4 subscales with good reliability (sadness-depression, anxiety, anger-hostility and happiness); the items range from 0 to 10 (0=nothing, 10=much).
Sleep quality. | Change from Baseline (at the beginning of the study) to 12 weeks (postintervention) and to 6 months (follow-up).
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), a validated questionnaire that includes 19 self-related questions ranging from 0 to 3. The total score ranges from 0 to 21, and a lower score indicates better quality of sleep.

OTHER OUTCOMES:
Safety and adverse events (AEs). | 12 weeks (postintervention)
  Safety will be assessed by the occurrence of any AEs using CTCAE version 5.0.
Satisfaction questionnaire. | 12 weeks (postintervention)
  Satisfaction will be registered by a questionnaire previously used in other clinical settings at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia Galiano-Castillo, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request. IPD that underlie the results reported in the future article/s, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Lozano-Lozano M, Lopez-Garzon M, Cuadrado-Guerrero P, Postigo-Martin P, Fernandez-Lao C, Tovar-Martin I, Galiano-Castillo N. Reliability of the electronic patient reported outcome measures for assessing xerostomia, dysphagia and quality of life in Spanish patients with head and neck cancer: a randomised crossover design. Health Qual Life Outcomes. 2025 Mar 3;23(1):19. doi: 10.1186/s12955-025-02347-1. PMID 40033397
- [Derived] Lopez-Garzon M, Lopez-Fernandez MD, Ruiz-Martinez AM, Galvan-Banqueri P, Lozano-Lozano M, Tovar-Martin I, Postigo-Martin P, Ariza-Vega P, Artacho-Cordon F, Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-Gualda MA, Arroyo-Morales M, Ruiz-Villaverde R, Galiano-Castillo N. Efficacy of photobiomodulation therapy combined with mobile health education in patients with head and neck cancer suffering from chronic xerostomia after radiotherapy: protocol for a three-arm, randomised, placebo-controlled, double-blinded study. BMJ Open. 2024 Jan 24;14(1):e078068. doi: 10.1136/bmjopen-2023-078068. PMID 38267245